CLINICAL TRIAL: NCT03846596
Title: Flow Cytometry Analysis of the Reactive Oxygen Species in Immature Granulocytes in Septic Patient
Acronym: SEPSIROS
Status: Terminated | Type: Observational
Why Stopped: Not enough patient
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18-0031 (SEPSIROS)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Sepsis
Keywords: Sepsis; reactive oxygen species; immature neutrophils
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Evaluated: An additional blood tube will be taken from patients hospitalized in intensive care or emergency department for acute sepsis
  Interventions: Biological: Additional blood tube

INTERVENTIONS:
Biological: Additional blood tube — Additional blood tube during care

SUMMARY:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. Early during sepsis course, immature neutrophils could be found in the bloodstream and may be less efficient than mature neutrophils in reactive oxygen species (ROS) production. ROS induce an oxidative stress for bacteria which can protect through the SOS response. The main objective is to evaluate the level of ROS produced in the early steps of sepsis by the immature neutrophils.

DETAILED DESCRIPTION:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. The immune system is activated by both pathogen-associated and host-derived molecular patterns. A strong response of neutrophils is engaged and both innate and adaptive immune system homeostasis are strongly affected. Neutrophils are able to produce high concentrations of inducible reactive oxygen species (ROS), leading to an oxidative stress. ROS can be released extracellularly at the site of infection or intracellularly in the phagolysosome. At early phase of sepsis, immature granulocytes are present in the bloodstream and could help to predict sepsis deterioration. However, it has also been shown that they are less efficient than mature granulocytes in ROS production and phagocytosis. ROS are potent stressors for bacteria and can directly or indirectly damage DNA. Bacteria can protect against DNA damage through the SOS response, which is a coordinated cellular response regulated by a repressor, LexA, and a sensor/activator, RecA. The bacterial SOS response is involved in acquisition of resistances to antibiotics through increasing frequencies of spontaneous mutations or increasing the expression of resistance and adaptation genes. The hypothesis that the low-level production of ROS by immature granulocytes in the early steps of sepsis could be beneficial for both the host, as a high level of ROS induce organ damage and dysfunction, and the pathogen, as low concentrations of ROS would be able to induce the SOS response allowing bacteria to enhance an adaptive response. The main objective it is to evaluate the level of ROS produced by the immature granulocytes in septic patient. Then, it will be assess if it could promote antibiotic resistance expression via SOS-induced integron gene cassette rearrangements.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients hospitalized in ICU or ED for acute sepsis

Exclusion Criteria:

* Immunosupressed patients
* Active cancer
* HIV
* Hematological or inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in intensive car or emergency department for acute sepsis
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
ROS level by Flow cytometry in immature granulocytes dosage sepsis | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the amount of ROS contained in the immature granulocytes from the onset of sepsis to the acute phase

SECONDARY OUTCOMES:
ROS level by Flow cytometry in mature granulocytes dosage sepsis | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the amount of ROS contained in the mature granulocytes from the onset of sepsis to the acute phase
Bacterial phagocytosis capacity of granulocytes assess by flow cytometry | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the number of ingested bacteria.
SOS response activation by bacteria determined by flow cytometry | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the expression of the SOS gene by the bacteria.
Hospital mortality | Day 28
  number of death
ROS level by Flow cytometry in monocyte dosage sepsis | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the amount of ROS contained in the monocyte from the onset of sepsis to the acute phase
ROS level by Flow cytometry in lymphocyte dosage sepsis | Day 1
  The biological variable obtained is an average of fluorescence intensity (MFI) corresponding to the amount of ROS contained in the lymphocyte from the onset of sepsis to the acute phase

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DAIX, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges university Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No